CLINICAL TRIAL: NCT01394107
Title: Evaluation of the Impact of the Thromboprophylactic Dose of LMWH on Coagulation in Pregnant Women.
Brief Title: Evaluation of the LMWH Thromboprophylaxis in Pregnancy
Status: Active, not recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Blaha, MD, PhD., M.D., PhD., Charles University, Czech Republic
Other Study IDs: LMWH_jB
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy
Keywords: Thromboprophylaxis; Effect of LMWH on coagulation; Pregnancy; Neuraxial anesthesia; Spinal haematoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant: 50 pregnant women with physiological ongoing pregnancy and undergoing planned caesarean section, without known coagulation disorders, will be included in to the study.
  Inclusion criteria: pregnant women undergoing planned caesarean section, 39th-40th week of pregnancy, age 18-40 years, informed consent.
- Control: 50 healthy women in fertility age (18-40 years) undergoing elective surgery for other than oncology or inflammatory indication, without known risk factors for coagulation disorders, not using hormonal contraception, informed consent.

SUMMARY:
The project aims to clarify the effect of the thromboprophylactic LMWH dose on coagulation in pregnant women just before birth, at the period of maximal physiological hypercoagulable state and with high risk of thromboembolism, the most common cause of maternal mortality in developed countries. Although LMWH are now routinely administered as prevention of thromboembolism, their effect on coagulation in pregnant women was not yet studied. The doses of LMWH in pregnancy are only derived in terms of coagulation from totally different groups of patients (surgical, orthopedic). We therefore will map the effect of thromboprophylactic LMWH dose on coagulation in pregnant women using recently available methods, especially a complex examination of coagulation within 24 h after LMWH application using thrombelastography, including examination with heparinase, and monitoring the effect of LMWH by measuring antiXa and TGT (thrombin generation time) activity. Based on these results we will also evaluate the possible influence of LMWH prophylaxis on the risk of spinal haematoma during neuraxial analgesia/anesthesia for delivery/Caesarean section. On the basis of our pilot results we can presume the current dosage of LMWH in pregnant women is inadequate and that it would be appropriate to adjust presently used dosage. At the same time we want to prove that the standard LMWH thromboprophylaxis in pregnant women does not increase the risk of spinal haematoma during neuraxial blockade. In both situations the targeted outcome is to increase the safety of pregnant women.

DETAILED DESCRIPTION:
AIMS OF THE PROJECT:

The aim of this project is to map the effect of the thromboprophylactic dose of LMWH on coagulation of women at the end of pregnancy, using recently available methods and laboratory tests, and simultaneously to evaluate the possible influence of LMWH on incidence of spinal hematoma. The methodology is based primarily on a complex examination of coagulation by thrombelastography (TEG), including comparative tests with heparinase, and on the monitoring effect of LMWH by measuring thrombin generation time (TGT) and levels of AntiXa. At the same time and, in cooperation with the Thrombotic Centre, standard and special laboratory hematology tests will be performed (INR, APTT, TT, fibrinogen, AT III, D-dimer, protein S, protein C, APC resistance, PFA, F VII, F VIII, PFA 100, TAT micro, vWf, APA, t-PA, PAI-1, blood count) together with genetic tests for FV Leiden and prothrombin II mutations.

HYPOTHESIS AND EXPECTED RESULTS:

We assume that with hypercoagulation and other influencing factors in pregnancy, the effect of LMWH on coagulation, compared to the population of non-pregnant women, will be significantly lower. Thus significantly lower will be also the effect of TED prophylaxis. For the same reason we assume that the current thromboprophylactic dosage of LMWH could not affect coagulation of pregnant women enough to increase the risk of spinal hematoma with neuraxial analgesia/anaesthesia administration.

SPECIFIC AIMS:

Primary aims: To map the coagulation effect of standard prophylactic dose of LMWH in pregnant women at the end of pregnancy. Based on these results, to evaluate the possible prophylactic effect of LMWH on TED prevention in pregnant compared to non-pregnant women and to evaluate the possible influence of LMWH on the potential risk of spinal hematoma development during neuraxial blockade in pregnancy.

Secondary aims: To propose a change of the thromboprophylactic regimen in pregnancy. To suggest a change of the recommended time interval between LMWH application and administration of neuraxial blockade in pregnant women.

METHODS AND RESEARCH SAMPLE CHARACTERISTICS:

Study design: prospective, monitoring

Size and type of study group: a total of 50 pregnant women with physiological ongoing pregnancy and undergoing planned caesarean section, without known coagulation disorders, will be included in to the study

Inclusion criteria: pregnant women undergoing planned caesarean section, 39th-40th week of pregnancy, age 18-40 years, informed consent.

Exclusion criteria: disapproval or non-cooperation of the mother, allergy to LMWH, coagulation disorders or the risk of, anticoagulant therapy in the last 3 months, signs of infection, history of cancer, signs of thrombosis or a history of thrombosis, the ongoing non-physiological pregnancy, significant obesity, or other severe comorbidity.

Withdrawal criteria: development of obstetric complications in the mother or foetus during the study following, finding of prothrombotic state.

Control group: 50 healthy women in fertility age (18-40 years) undergoing elective surgery for other than oncology or inflammatory indication, without known risk factors for coagulation disorders, not using hormonal contraception, informed consent.

LMWH applications: a standard thromboprophylactic dose of LMWH (4000 IU of enoxaparin subcutaneously) will be given to pregnant woman/patient in control group.

Monitoring of coagulation: To evaluate coagulation changes after administration of LMWH dose we will perform thrombelastographic examination (TEG; Haemascope Corp., USA.) of venous blood (including examination with heparinase) and specific laboratory tests to measure the effect of LMWH activity - antiXa and TGT (thrombin generation time). Coagulation system will be also be examined by other available laboratory tests (INR, APTT, TT, fibrinogen, AT III, D-dimer, protein S, protein C, APC resistance, PFA, F VII, F VIII, PFA 100, TAT micro, vWf, APA, t-PA, PAI-1, blood count) including genetic testing for FV Leiden and prothrombin II mutation.

Monitoring of coagulation takes place in four phases:

1. Basal level - before LMWH application
2. The maximum effect of LMWH - 4 hours after application
3. Low efficiency of LMWH - 8 hours after application
4. Control level of LMWH effectiveness - 24 hours after application

Samplings for laboratory testing will be performed in the same way as a sample for TEG examination - venous blood will be in planned times taken by one-time blood draw to prevent premature coagulation activation and dilution of the sample. Blood samples will be collected according to standard guidelines (for coagulation tests and TEG in a test tubes with sodium citrate) - and subsequently processed in Central haematology laboratory.

For TEG examination 1 ml of whole blood will be activated by 1% celite and then 360 μl of sample (340 μl blood + 20 μl CaCl2) will be analyzed in a standard cuvette and 360 μl of sample (340 μl blood + 20 μl CaCl2) in the cuvette with heparinase. Following parameters will be recorded: time r, time K, angle alpha, maximum amplitude MA and LY30 as a factor of fibrinolysis. From the measured values coagulation index (CI) will be calculated.

DATA COLLECTION:

Demographic, obstetric and clinical data - age, height, weight, BMI, gestational age, previous pregnancy, associated medical conditions. Standard pre-operative assessment and pharmacological history. Fluid intake and output during the surveillance. Any bleeding and / or thromboembolic complications from beginning of the study to the end of hospitalization after Cesarean section.

DATA PROCESSING:

All data will be stored at electronic database with safety back up. Statistical analysis will be performed in cooperation with Biomedical Statistics Dept. of the Institute of Biophysics and Informatics, Charles University in Prague, 1st Faculty of Medicine. Based on preliminary analysis the overall number of subjects was determined as 50 in both study groups.

DATA EVALUATION:

Based on study results the relationship between the potential risk of spinal hematoma and the LMWH application will be evaluated by the Expert Committee for Obstetric Anaesthesia of the Czech Society of Anaesthesiology and Intensive Care Medicine (ČCSARIM). The conclusions and the resulting recommendations will be submitted to the Executive Committee of ČSARIM.

TIME SCHEDULE:

Based on the feasibility test and pilot study we consider as real inclusion 3 patients into the study per month. This number is based on the number of anticipated elective caesarean operations and the possibility of recruiting appropriate subjects satisfying all the criteria, and also on organizational difficulties when samples at study hour 8 and 24 will be taken at the place of subject's residence.

1. st year - creating a study database, patient recruitment, inclusion of 15 pregnant women + 15 controls; samples processing.
2. nd year - recruiting patients, inclusion of 25 pregnant women + 15 controls, processing and analysis of samples, evaluation and presentation of preliminary study data.
3. rd year - recruiting patients, inclusion 10 pregnant women + 20 controls, processing and analysis of samples. The evaluation of all study data, statistical evaluation, presentation and publication the final results.

DEPARTMENTS INVOLVED, PRINCIPAL INVESTIGATOR´S READINESS:

Department of Anaesthesiology and Intensive Care Institute of Clinical Biochemistry and Laboratory Diagnostics, Central Hematology Laboratory, Thrombotic Centre Department of Gynaecology and Obstetrics

EXPECTED RESULTS AND PROJECT IMPORTANCE:

The expected project outcome is the detailed evaluation of the influence of LMWH on coagulation in pregnant women and suggested modification of dosing schemes for thromboprophylaxis before Caesarean operation, which would better reflect physiological hypercoagulation in pregnancy. Due to improved TED prophylaxis the main long-term outcome then should be the reduction of maternal mortality in connection to thromboembolic diseases. At the same time we want to prove that the current dosage of LMWH in pregnant women cannot increase the risk of epidural hematoma during neuraxial blockades and we would recommend changes of time relationships between administration of LMWH and neuraxial blockade.

COOPERATION ON THE PROJECT:

The project will be performed in cooperation between the Dept. of Anaesthesiology and Intensive Care, Thrombotic Centre of Institute of Clinical Biochemistry and Laboratory Diagnostics and Dept. of Gynaecology and Obstetrics.

The relationship between the risk of spinal hematoma and the LMWH applications will be evaluated by the Expert Committee for Obstetric Anaesthesia and Executive Committee of the Czech Society of Anaesthesiology and Intensive Care Medicine.

DISCUSSION:

So far, no studies have been published dealing with the influence of thromboprophylactic LMWH dose on coagulation in pregnant women. The only study, showing a reduced effect of LMWH during pregnancy, was only evaluating its effect on antiXa activity. Our project differs in complexity and range of other available methods used such as thrombin generation time and especially thrombelastography. Thus our project also builds on the results of previous grant project IGA No. NR8157 "The use of thrombelastography in evaluating coagulation in women with physiologically and pathologically ongoing pregnancy, during birth and beyond".

EXPECTED PROJECT BENEFITS AND IMPACTS OF THE PROPOSED PROJECT The project aims to clarify the effect of LMWH on coagulation in pregnant women just before birth, at a period of maximal physiological hypercoagulable state and with high risk of thromboembolism, the most common cause of maternal mortality in developed countries. Although LMWH are now routinely administered as prevention of thromboembolism in all women undergoing Caesarean operation, their effect on coagulation in pregnant women was not yet studied. Research of haemocoagulation in pregnant women worldwide is rather difficult, so the results of such a project are highly awaited and are then a great opportunity to present Czech research on European and World forums.

The main expected benefit of this project will be the evaluation of the adequacy of current LMWH thromboprophylaxis in pregnant women (which is recently only derived from surgical patients). The next important study outcome will be the evaluation of possible influence of the LMWH thromboprophylaxis on risk of spinal hematoma in connection to neuraxial anaesthesiology techniques in pregnant women. In both situations the targeted outcome is to change present recommendations to increase the safety of pregnant women undergoing Caesarean operation. Just in Czechia this issue affects about 30 000 women/year.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women undergoing planned caesarean section
* 39th-40th week of pregnancy
* age 18-40 years

Exclusion Criteria:

* disapproval or non-cooperation of the mother
* allergy to LMWH
* coagulation disorders or the risk of
* anticoagulant therapy in the last 3 months
* signs of infection
* history of cancer
* signs of thrombosis or a history of thrombosis
* the ongoing non-physiological pregnancy
* significant obesity, or other severe comorbidity

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women undergoing planned caesarean section, 39th-40th week of pregnancy, age 18-40 years
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Effect of standard prophylactic dose of LMWH on coagulation in pregnant women | 24 hours after LMWH application
  To map the coagulation effect of standard prophylactic dose of LMWH in pregnant women at the end of pregnancy. Based on these results, to evaluate the possible prophylactic effect of LMWH on TED prevention in pregnant compared to non-pregnant women.

SECONDARY OUTCOMES:
Evaluation of the possible influence of LMWH on the potential risk of spinal hematoma development during neuraxial blockade in pregnancy. | 24 hours after LMWH application

CONTACTS AND LOCATIONS:
Overall Officials: Jan Blaha, MD, PhD, Principal Investigator — Charles University, 1st Medical Faculty in Prague
Locations (1):
- General University Hospital in Prague, Prague, Czechia